CLINICAL TRIAL: NCT06988995
Title: Compassion Strikes Back: Improving Dyadic Quality of Life for LVAD Patients and Caregivers
Brief Title: Compassion Strikes Back
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202500512
Record Dates: First submitted 2025-05-05; First posted 2025-05-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-05

CONDITIONS: LVAD Caregivers; LVAD (Left Ventricular Assist Device); Quality of Life (QOL); Self-Compassion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meeting (Experimental)
  Interventions: Behavioral: Meeting
- Information (Active Comparator)
  Interventions: Other: Information

INTERVENTIONS:
Other: Information — Participants provided handouts with information on self-compassion
  Arms: Information
Behavioral: Meeting — Participants meet with a psychological provider to receive information on self-compassion and training on how to utilize self-compassion
  Arms: Meeting

SUMMARY:
Research has shown that LVAD patients and their caregivers typically experience increased mental health concerns and decreased quality of life following LVAD implantation and hospital discharge. The purpose of this study is to explore how to improve quality of life for LVAD patients and their caregivers in the initial transition from hospital to home after LVAD implantation.

Over the course of the study, participants will complete 2 surveys: one when participants are in the hospital and one at a 2-month post-hospital follow-up appointment with the participants' cardiologist. Participants may be contacted if there is data missing from surveys.

Participants may also be provided with information on improving mental health in the form of handouts or a brief meeting with a psychology provider.

ELIGIBILITY:
Inclusion Criteria:

* LVAD implantation or caregiver or patient with LVAD; over 18 years old; primary caregiver is a family member

Exclusion Criteria:

* Currently or in the past 3 months received psychotherapy or psychosocial or peer support; hospitalized for psychiatric reasons in the past 6 months; current, active suicidal thoughts or a reported suicide attempt within the past year; a current alcohol/substance use disorder that required immediate treatment; or a current or past thought disorder, psychosis, or unmanaged bipolar disorder; enrolled in another investigational research/clinical trial; toxic/negative dynamic between pt and caregiver; extended post-LVAD implantation course (i.e., more than 2 months in the hospital).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Self-compassion | 2 months
  Level of self-compassion a participant reports using the Self-Compassion Scale - Short Form (Raes et al., 2011). Scores range from 1-5.
QOL | 2 months
  Quality of Life will be measured using the 16 item Quality of Life Scale (Burckhardt et al., 1989). Scores range from 16-112, with higher scores indicating higher levels of quality of life.

SECONDARY OUTCOMES:
NYHA | 2 months
Cardiac Self-Efficacy | 2 months
  The Cardiac Self-Efficacy Scale (Sullivan et al., 1998) is a 13-item measure that measures self-efficacy in patients with cardiac problems across 2 subscales: maintain and control. Scores are averaged across the two subscales. Scores range from 0-4, with higher scores indicating higher confidence or perceived self-efficacy.
General Self-Efficacy | 2 months
  General Self-efficacy will be measured by the General Self-Efficacy Scale (Weinman et al., 1995). The GSE is a 10-item scale with scores ranging from 10-40, with higher scores indicating more self-efficacy.
Illness Denial | 2 months
  Illness denial will be measured using the Illness Denial Questionnaire. Caregivers will receive the caregiver version, and patients will receive the patient version. Both versions are 24-items, with scores ranging from 0-24. Higher scores indicate higher levels of denial
Perceived Stress Scale | 2 months
Caregiver Burden | 2 months
  Caregiver burden will be assessed using the Zarit Burden Interview - Short Form, which is a 12 item questionnaire assessing caregiver burden. Scores range from 0-48, with a score over 20 indicating high burden.
Acceptability & Feasibility of Intervention | 2 months
  Participants will be asked about the feasibility and acceptability of the intervention they receive. Scores range from 0-5, with higher scores indicating greater acceptability and higher feasibility (i.e., the intervention felt easy to complete and use).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No